CLINICAL TRIAL: NCT03455127
Title: Community Based Lay Worker Pilot of FSI-ECD
Brief Title: Alliance for Family Strengthening: Improved Early Childhood Development in Rwanda
Acronym: FSI-ECD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: World Bank (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Network of European Foundations (Unknown); The ELMA Foundation (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-16 1570_Activity B
Record Dates: First submitted 2017-11-09; First posted 2018-03-06 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Child Development
Keywords: Child Development; Home Visiting; Parenting Program; Social Protection; Public Works

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic Public Works as Usual (No Intervention): Half of the sample will be eligible to receive or be receiving the Government of Rwanda's (GOR) flagship social protection programming, Vision 2020 Program (VUP). One component of this program is to provide cash for work opportunities for labor endowed vulnerable households, i.e. one able bodied adult. Vulnerable households are those in Poverty Level 1 category, the GOR's poverty classification system. Furthermore, this study will require households in the control group receiving classic public works as usual to have at least one child between the ages of 6 months to 36 months.
- Classic Public Works + FSI ECD (Experimental): Half of the sample will receive the FSI ECD home visiting parenting program alongside the GOR's classic public works programming. These households will be in Poverty Level 1 with an able-bodied adult, thus eligible to receive or be received the GORs public works programming. They will have a child between 6 and 36 months at enrollment. Households will be visited by a trained community based lay worker on a weekly to biweekly basis to deliver the 15 module curriculum covering a range of topics from nutrition, water and sanitation, hygiene, early stimulation, conflict management, to good communication. The intervention seeks to promote healthy child development via active coaching to individual beneficiary households, delivering modules on a one on one basis and engaging all family members.
  Interventions: Other: FSI ECD

INTERVENTIONS:
Other: FSI ECD — Households will be visited by a trained community based lay worker on a weekly to biweekly basis to deliver the 15 module curriculum covering a range of topics from nutrition, water and sanitation, hygiene, early stimulation, conflict management, to good communication. The intervention seeks to promote healthy child development via active coaching to individual beneficiary households, delivering modules on a one on one basis and engaging all family members.
  Other Names: Family Strengthening Intervention for ECD
  Arms: Classic Public Works + FSI ECD

SUMMARY:
Preliminary pilot testing of the home-based FSI-ECD intervention as delivered by community based lay workers.

DETAILED DESCRIPTION:
The Family Strengthening Intervention for early childhood development was created and piloted for feasibility and acceptability in an ongoing protocol #15440 with Harvard Internal Review Board titled, "Developing and Piloting a Quantitative Behavioral Assessment Battery, Estimating Prevalence of Mental Disability among HIV/AIDS-affected Youth, and Piloting an Adapted Mental Health Intervention for HIV/AIDS-Affected Children in Rwanda." Research personnel have been adapting the existing recruitment materials/sessions and 15 Module Manual (FSI-ECD) with a focus on making the manual and corresponding materials more user friendly for community based lay worker "coaches."

This preliminary testing will provide an opportunity to administer a planned full scale 1,000+ household cluster randomized control trial on a smaller scale in order to learn from our materials that have been adapted for community based lay workers. This will also allow us to test our supervision and training structures to make necessary adaptation ahead of the planned full scale trial.

After all beneficiary households have completed the FSI-ECD intervention, each community based lay worker will complete a qualitative and quantitative exit assessment of his/her experience delivering the intervention, as well as ongoing feedback during the administration of FSI-ECD; allowing for the intervention and support structure to be strengthened for future iterations.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiary Inclusion Criteria: All participants must live in chosen District(s) of Rwanda. Inclusion criteria for families are: (a) being VUP-eligible, (b) having at least one children aged 6-36 months living in the home and (c) having caregiver willing to discuss and enhance their parenting practices by interacting with a home-visiting coach. Caregiver eligibility: (a) is aged 18 or older and cares for child(ren) and (b) lives in the same household as child(ren). We will enroll both single and dual caregiver families to reflect population dynamics. Legal guardians may be aunts, uncles, grandparents, or foster parents.

Community Based Lay Worker Exclusion Criteria: Community based workers selected to deliver the FSI-ECD intervention must: (a) live in the sector of beneficiary households they will deliver the intervention to, (b) be Rwanda, (c) be aged 18 or older; (d) be able to write, read, and count in local language; (e) be committed to young children and family values; (f) have the required amount of time to carry out the FSI-ECD intervention with a select number of households, (e) be recommended and approved by local community and authorities.

Exclusion Criteria:

* Beneficiary Exclusion Criteria: Potential participants will be excluded if they do not live in chosen District of Rwanda, do not have children between the ages of 6 and 36 months living in their household for whom they are the primary caregiver, they are not eligible/enrolled in Rwanda's public works social protection program, VUP, or have severe cognitive impairments which preclude their ability to speak to the research questions under study. We will exclude families in the midst of crisis (e.g., a caregiver with active suicidal attempts or psychosis) and refer them to appropriate services.

Community Based Lay Worker Exclusion Criteria: Community based workers will not be selected to deliver the FSI-ECD intervention if they do/are not: (a) live in the sector of beneficiary households they will deliver the intervention to, (b) Rwanda, (c) aged 18 or older; (d) able to write, read, and count in local language; (e) committed to young children and family values; (f) have required amount of time to carry out the FSI-ECD intervention with a select number of households, (e) recommended and approved by local community and authorities.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Ages Stages Questionnaire-3 | 12 months/18 months
  Change in Child Communication, Fine Motor, Gross Motor, Problem Solving, and Personal Social Development

SECONDARY OUTCOMES:
Hopkins Symptoms Check List | 12 months/18 months
  Change in Caregiver Mental Health
Multiple Indicator Cluster Survey 5 | 12 months/18 months
  Change in Infant and Young Child Feeding Practices
Rwanda Comprehensive Food Security and Vulnerability Analysis and Nutrition Survey | 12 months/18 months
  Change in Assessing Household Food Security related to diversity of food and meal frequency
Local Derived Scale | 12 months/18 months
  Change in Family Trust and Unity
System for Observing Family Therapy Alliances | 12 months
  Interventionist Self-Report
Difficulties in Emotional Regulation (DERS) | 12 months/18 months
  Change in Caregiver Emotional Regulation
Malawi Development Assessment Tool (MDAT) | 12 months/18 months
  Change in Child Development Observational Measure for Fine Motor, Gross Motor and Language
Home Observation for the Measurement of the Environment (HOME Inventory) | 12 months/18 months
  Change in Home Environment
Observation of Mother Child Interaction (OMCI) | 12 months/18 months
  Change in Caregiver-Child Relationship/Stimulation
Ages Stages Questionnaire Socio-Emotional | 12 months/18 months
  Change in Child Socio-Emotional Development

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, Sc.D., M.A., Principal Investigator — Boston College School of Social Work
Locations (1):
- Rwamagana District, Rubona, Rwanda